CLINICAL TRIAL: NCT02823886
Title: Inflammatory Response in Myocardial Infarction Evaluated by MRI and Biomarkers of Inflammation
Brief Title: Inflammatory Response in Myocardial Infarction Evaluated by MRI and Biomarkers
Acronym: RIFIFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL16_0130
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; MRI; inflammatory biomarkers
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STEMI patients (Experimental)
  Interventions: Other: MRI at D7; Biological: Blood samples

INTERVENTIONS:
Other: MRI at D7 — The infarct size measured on MRI at 7 days.
Biological: Blood samples — Blood samples at H0; H4; H12; H24, H48, D7 and 1 month post MI

SUMMARY:
An intense inflammatory reaction is triggered by the ischemic injury during myocardial infarction. The inflammatory processes involved are complex and haven't been explored in detail in human patients. This inflammatory response can increase myocardial damage following reperfusion, leading to adverse remodeling and adverse events (heart failure, sudden cardiac death).

Cardiac MRI can assess the size of myocardial infarction and many other parameters associated with myocardial injury: edema, hemorrhage, micro-vascular obstruction.

(However the association between biomarkers of inflammation and these imaging parameters is not known).

There is very little data correlating imaging markers of myocardial injury to the biokinetics of inflammation biomarkers.

In this study, the aim is to assess the relationship between the kinetics of specific inflammatory biomarkers (interleukin-1beta, interleukin 6, interleukin 17, Tumor Necrosis Factor (TNF)-alpha, C reactive protein (CRP), soluble toll-like receptor-2 (ST2), neutrophils) and imaging markers of injury measured by cardiac MRI at the acute phase in 20 acute mycardial infarction (AMI) patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients, aged over 18, without any legal protection measure,
* Having a health coverage,
* Presenting within 12 hours of the onset of chest pain,
* Who have ST segment elevation ≥0.2 millivolt (mV) in two contiguous leads,
* For whom the clinical decision was made to treat with percutaneous coronary intervention (PCI).
* he culprit coronary artery has to be the left anterior descending (LAD) or the right coronary (RC)
* The LAD or RC artery has to be occluded (TIMI flow grade 0-1) at the time of admission coronary angiography.
* Preliminary oral informed consent followed by signed informed consent as soon as possible
* Final TIMI ≥ 2

Exclusion Criteria:

* Female patients currently pregnant or women of childbearing age who were not using contraception (oral diagnosis).
* Patients with cardiogenic shock
* Patient in Cardiac arrest
* History of Myocardial Infarction
* Contre-indication to MRI : claustrophobia, pacemaker or cardiac defibrillator , eye metal body allergy to gadolinium
* Patient with Atrial Fibrillation.
* Patients with loss of consciousness or (Glasgow <14)
* known renal insufficiency (either known creatinin clearance < 30 ml/min/1.73m² or current medical care for severe renal insufficiency)
* Patients with any disorder associated with immunological dysfunction
* Adult with legal protection measure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Relationship between interleukin-1beta serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between interleukin 6 serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between interleukin 17 serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between TNF-alpha serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between CRP serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between ST2 serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days
Relationship between polymorphonuclear neutrophil serum level and infarct size | Day 7
  the relationship between serum measured at H24 and the infarct size measured on MRI at 7 days

SECONDARY OUTCOMES:
Relationship between H24 peak or area under curve interleukin-1beta serum level and the size of no reflow | Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve interleukin 6 serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve interleukin 17 serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve TNF-alpha serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  and concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve CRP serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  and concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve polymorphonuclear neutrophil serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  and concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
Relationship between H24 peak or area under curve ST2 serum level and the size of no reflow | Hour 24, Hour 48, Day 7 and 1 month post MI for biomarkers and Day 7 for the MRI
  concerning the MRI, it is the measure of myocardial oedema, intracardiac hemorrhage and microvascular obstruction measured on MRI
relationship between the H24 peak values of serum level for interleukin 1 beta and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for interleukin 6 and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for interleukin 17 and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for TNF-alpha and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for CRP and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for ST2 and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for polynuclear neutrophil and the cardiovascular events | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day7 and 1 month post MI) for biomarkers and follow up at 1 month
relationship between the H24 peak values of serum level for interleukin-1beta and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.
relationship between the H24 peak values of serum level for interleukin 6 and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.
relationship between the H24 peak values of serum level for interleukin 17 and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.
relationship between the H24 peak values of serum level for TNF-alpha and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.
relationship between the H24 peak values of serum level for CRP and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.
relationship between the H24 peak values of serum level for ST2 and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days..
relationship between the H24 peak values of serum level for polymorphonuclear neutrophil and functional and anatomical parameters | area under curve (pharmacokinetic : Hour 0; Hour 4; Hour 12; Hour 24, Hour 48, Day 7 and 1 month post MI) for biomarkers and D7 for the MRI
  relationship between area under curve and functional and anatomical parameters (end-systolic volume and end -diastolic Volume) measured on MRI at 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] This study confirms the strong association between infarct size and CRP levels, but does not demonstrate any significant relationship with the other biomarkers investigated (IL-6, IL-8, and IL-10). Among the three markers of myocardial injury assessed, myocardial hemorrhage appears to be strongly associated with the release of inflammatory biomarkers following reperfused STEMI. Attenuation of reperfusion-induced hemorrhage may therefore represent a novel therapeutic target for future adjunctive treatments in STEMI patients. Additional cytokine measurements are currently being performed to further refine the assessment of the relationship between hemorrhage, infarct size, and other inflammatory biomarkers.